CLINICAL TRIAL: NCT03250728
Title: Role of the Endothelium in Stroke-like Episode Among CDG Patients
Acronym: PECDG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: K170703J; 2017-A02141-52 (Registry Identifier: ANSM-IDRCB)
Record Dates: First submitted 2017-08-11; First posted 2017-08-16 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Congenital Disorders of Glycosylation
Keywords: CDG; Stroke-like; Endothelial progenitor cells (EPCs); Protein C; Congenital Disorders og Glycosylation
MeSH Terms: conditions — Congenital Disorders of Glycosylation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CDG with stroke-like history (Other)
  Interventions: Biological: Peripheral blood puncture
- CDG without stroke-like history (Other)
  Interventions: Biological: Peripheral blood puncture

INTERVENTIONS:
Biological: Peripheral blood puncture — Endothelial progenitor cells will be isolated from peripheral blood by density gradient and cultured in 10%FBS EGM2 medium
  On the EPCs we will study:
  * the endothelial permeability
  * the protein C system

SUMMARY:
The aim of the study is to evaluate the role of the endothelial barrier in the occurrence of stroke-like episode. And to study the protein C system on the surface of the endothelium.

DETAILED DESCRIPTION:
The study consists in isolating endothelial progenitor cells in peripheral blood. After blood puncture, PBMC (peripheral blood mononuclear cell) are isolated by Ficoll gradient and then culturing in appropriated medium.

When cells are confluent, investigators can study the endothelial barrier by using permeability assay and transendothelial resistance test (iCELLigence technology).

Then, protein C system will be studied. Indeed, EPCR (Endothelial protein C receptor) and TM (thrombomodulin), are the two receptors responsible for the activation of protein C. The expression of these receptors will be assessed in flow cytometry. The activated protein C is able to interact with the third receptor PAR1 (Protease activated receptor 1) which is responsible for the protective effects of the on the endothelial barrier. The PAR1 expression will be studied in flow cytometry also.

In order to measure the capacity of the protein C system to generate activated protein C investigators will assay an activated protein C generation on the cell surface.

All these assays will be realized in basal condition and in heat stress (42°C), to mimic the stroke-like episode environment. Indeed, stroke-like episodes occur always during febrile illness.

ELIGIBILITY:
Inclusion Criteria:

* patients with CDG molecularly diagnosed
* with stroke-like history or not

Exclusion Criteria:

* rejection to participate in research

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-11-23 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-04-26 (Actual)

PRIMARY OUTCOMES:
Endothelial permeability assay in basal condition | at inclusion
Endothelial permeability assay after an heat shock | at inclusion

SECONDARY OUTCOMES:
Activated protein C generation assay on the endothelial cell surface | at inclusion
Quantification of the endothelial receptors (EPCR, TM, PAR1) | at inclusion
Endothelial permeability assay after an activated protein C incubation | at inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Pascale De Lonlay, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Delphine Borgel, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Necker enfants malades, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No